CLINICAL TRIAL: NCT05941767
Title: Comparing Intravenous Versus Nebulized Either Lidocaine or Dexmedetomidine for Attenuation of the Hemodynamic Responses to Laryngoscopy and Intubation
Brief Title: Dexmedetomidine or Lidocaine for Lessening the Hemodynamic Responses to Laryngoscopy and Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Stress Response to intubation
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Anesthesia Intubation Complication
Keywords: Dexmedetomidine; Lidocaine
MeSH Terms: interventions — Dexmedetomidine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dexmedetomidine nebulization (Active Comparator): The patient will receive nebulized dexmedetomidine via face mask nebulizer (1mcg/kg) 20 minutes before induction.
  Interventions: Drug: Dexmedetomidine nebulization
- Lidocaine Nebulization (Active Comparator): The patient will receive nebulized lidocaine 4% (3 mg /kg) added to 2 ml normal saline 0.9% 10 minutes before induction of general anesthesia.
  Interventions: Drug: Lidocaine nebulization
- Dexmedetomidine IV (Active Comparator): The patient will receive an intravenous infusion of dexmedetomidine (1 ml= 4 mcg) via a syringe pump and will be started at a dose of 1 mcg/kg 20 minutes before induction of general anesthesia.
  Interventions: Drug: Dexmedetomidine IV
- Lidocaine IV (Active Comparator): The patient will receive 1.5mg/kg intravenous lidocaine 2% completed to 10 ml with normal saline 0.9% intravenous 90 seconds before induction of general anesthesia.
  Interventions: Drug: Lidocaine IV

INTERVENTIONS:
Drug: Dexmedetomidine nebulization — The patient will receive nebulized dexmedetomidine via face mask nebulizer 10 minutes before induction of general anesthesia.
  Other Names: Precedex (200 mcg/2ml)
  Arms: Dexmedetomidine nebulization
Drug: Lidocaine nebulization — The patient will receive nebulized lidocaine 4% (3 mg /kg) 10 minutes before induction of general anesthesia.
  Other Names: Lidocaine 2% (20 mg/ml)
  Arms: Lidocaine Nebulization
Drug: Dexmedetomidine IV — The patient will receive intravenous infusion via a syringe pump of dexmedetomidine (1 ml= 4mcg) started at a dose of 1 mcg/kg 20 minutes before induction of general anesthesia.
  Other Names: Precedex
  Arms: Dexmedetomidine IV
Drug: Lidocaine IV — The patient will receive 1.5 mg/kg lidocaine 2% (1 ml = 20mg) completed to 10 ml with normal saline 0.9% intravenous 90 seconds before induction of general anesthesia.
  Other Names: Lidocaine 2% (20 mg/ml)
  Arms: Lidocaine IV

SUMMARY:
Laryngoscopy, tracheal intubation, surgical stimulation, and extubation unleash remarkable sympathetic activity and are associated with transient but significant hemodynamic changes. The need to blunt these noxious responses effectively has led to using several techniques and pharmacological agents, local anesthetics, beta-adrenergic-blockers, calcium channel antagonists, and opioids with varied success. This study aims to evaluate the effect of nebulized and intravenous either dexmedetomidine or lidocaine for attenuating the hemodynamic responses to laryngoscopy and intubation.

DETAILED DESCRIPTION:
Hemodynamic responses to laryngoscopy and intubation are a significant concern for the anesthesiologist. Laryngoscopy, tracheal intubation, surgical stimulation, and extubation unleash remarkable sympathetic activity and are associated with transient but significant hemodynamic changes. These hemodynamic derangements can be lethal in patients with multiple comorbidities. The need to blunt these noxious responses effectively has led to using several techniques and pharmacological agents, local anesthetics, beta-adrenergic-blockers, calcium channel antagonists, and opioids with varied success. This study aims to evaluate the effect of nebulized and intravenous either dexmedetomidine or lidocaine for attenuating the hemodynamic responses to laryngoscopy and intubation.

ELIGIBILITY:
Inclusion Criteria:

* The American Society of Anesthesiologists (ASA) physical status I & II. BMI: ((≤ 35 kg/m2)). The patients are to be scheduled to undergo elective surgery under general anesthesia.

Mallampati grade I, II

Exclusion Criteria:

* Uncooperative patient. History of allergy to study drugs. Hemodynamically unstable patient. Renal or hepatic dysfunction or hypertensive patients.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2023-11-05 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
Change in serum cortisol levels. | Measurement will be done 45 minutes preoperative and 10 minutes after endotracheal intubation.
  Base line blood sample will be drawn 45 minutes preoperative and 10 minutes post intubation for cortisol level measurements.
Change in mean arterial blood pressure (MAP) in mmHg. | Measurement will be done 10 minutes before induction and at 1,3,5,7 and 10 minutes after endotracheal intubation.
  Mean arterial pressure (MAP) will be recorded 10 minutes before induction and at 1,3,5,7 and10 minutes after endotracheal intubation.
Change in heart rate (HR) per minute. | Measurement will be done 10 minutes before induction and at 1,3,5,7 and 10 minutes after endotracheal intubation.
  Heart rate (HR) will be recorded 10 minutes before induction and at 1,3,5,7 and10 minutes after endotracheal intubation.
Change in systolic blood pressure (SBP) in mmHg. | Measurement will be done 10 minutes before induction and at 1,3,5,7 and 10 minutes after endotracheal intubation.
  Systolic blood pressure (SBP)will be recorded 10 minutes before induction and at 1,3,5,7 and10 minutes after endotracheal intubation.
Change in diastolic blood pressure (DBP) in mmHg. | Measurement will be done 10 minutes before induction and at 1,3,5,7 and10 minutes after endotracheal intubation.
  Diastolic blood pressure (SBP)will be recorded 10 minutes before induction and at 1,3,5,7 and 10 minutes after endotracheal intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Zaki Saleh Taha, MD, Principal Investigator — Professor of Anesthesia, Intensive Care and pain management; Yasser Mohamed Nasr, MD, Principal Investigator — Professor of Anesthesia, Intensive Care and pain management
Locations (1):
- Faculty of medicine, Zagazig University, Zagazig, Al-Sharkia, Egypt

REFERENCES:
- [Background] Sriramka B, Warsi ZH, Sahoo J. Effects of adding dexmedetomidine to nebulized lidocaine on control of hemodynamic responses to laryngoscopy and intubation: A randomized clinical trial. J Anaesthesiol Clin Pharmacol. 2023 Jan-Mar;39(1):11-17. doi: 10.4103/joacp.JOACP_93_21. Epub 2022 Feb 10. PMID 37250266
- [Background] Misra S, Behera BK, Mitra JK, Sahoo AK, Jena SS, Srinivasan A. Effect of preoperative dexmedetomidine nebulization on the hemodynamic response to laryngoscopy and intubation: a randomized control trial. Korean J Anesthesiol. 2021 Apr;74(2):150-157. doi: 10.4097/kja.20153. Epub 2020 May 20. PMID 32434291
- [Background] Mahajan L, Kaur M, Gupta R, Aujla KS, Singh A, Kaur A. Attenuation of the pressor responses to laryngoscopy and endotracheal intubation with intravenous dexmedetomidine versus magnesium sulphate under bispectral index-controlled anaesthesia: A placebo-controlled prospective randomised trial. Indian J Anaesth. 2018 May;62(5):337-343. doi: 10.4103/ija.IJA_1_18. PMID 29910490
- [Background] Soltani Mohammadi S, Maziar A, Saliminia A. Comparing Clonidine and Lidocaine on Attenuation of Hemodynamic Responses to Laryngoscopy and Tracheal Intubation in Controlled Hypertensive Patients: A Randomized, Double-Blinded Clinical Trial. Anesth Pain Med. 2016 Mar 27;6(2):e34271. doi: 10.5812/aapm.34271. eCollection 2016 Apr. PMID 27247914
- [Background] Mahjoubifard M, Heidari M, Dahmardeh M, Mirtajani SB, Jahangirifard A. Comparison of Dexmedetomidine, Lidocaine, and Fentanyl in Attenuation Hemodynamic Response of Laryngoscopy and Intubation in Patients Undergoing Cardiac Surgery. Anesthesiol Res Pract. 2020 Jul 1;2020:4814037. doi: 10.1155/2020/4814037. eCollection 2020. PMID 32695159